CLINICAL TRIAL: NCT03155750
Title: Effects of Zero-Time Exercise (ZTEx) on Inactive Adults With Insomnia: A Pilot Randomized Controlled Trial
Brief Title: Effects of Zero-Time Exercise (ZTEx) on Inactive Adults With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, YEUNG Wing Fai, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZTEInsomnia
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Insomnia, Primary
Keywords: insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero Time Exercise training (Experimental): Subjects in this group will attend two 2-hour ZTEx training lessons. Each subject will receive a handout and an exercise log. The handout includes a picture-illustrating ZTEx step-by-step protocol. The exercise log is for them to record their time spending on performing the ZTEx every day during the 8-week study period.
  Interventions: Other: Zero Time Exercise
- sleep hygiene education (Active Comparator): Subjects in this group will receive two 2-hour lessons of sleep hygiene education delivered by a registered nurse.
  Interventions: Other: Sleep hygiene education

INTERVENTIONS:
Other: Zero Time Exercise — Zero Time Exercise encourage people to increase physical exercise by simple movements that can be done any time at any places. We offer a 2-session training course to train the subjects to do zero-time exercise.
  Arms: Zero Time Exercise training
Other: Sleep hygiene education — We offer a 2-session education course to teach the subjects about sleep hygiene practice.
  Arms: sleep hygiene education

SUMMARY:
Objectives: To evaluate the clinical effects of Zero-Time Exercise (ZTEx) for treating insomnia disorder delivered by a training course.

Hypothesis: Subjects in the ZTEx training group will have greater improvement in insomnia symptoms and daytime impairment than those in the sleep hygiene education (SHE) group at week 8.

Design and subjects: A randomized controlled trial. 32 inactive subjects with insomnia disorder recruited from the community will be randomized to ZTEx training or SHE groups in a 1: 1 ratio.

Study instrument: Insomnia Severity Index (ISI) will be used to assess insomnia symptoms and daytime impairment.

Interventions: Subjects in the ZTEx training group will attend two training lessons (2-hour each) to learn ZTEx and practice it every night for 8 weeks; subjects in the SHE group will receive sleep hygiene education with the schedule and duration that are same to the ZTEx training group.

Main outcome measures: The primary outcome measure is the ISI score. Other measures include sleep parameters by subjective sleep diary and objective actigraphy, Hospital Anxiety and Depression Scale, Multidimensional Fatigue Inventory-20 and Short Form-6 Dimension. Acceptability and compliance of ZTEx will be evaluated.

Data Analysis: Differences in the questionnaire scores, subjective and objective sleep parameters will be examined using a mixed-effects model.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-65 years old;
* Chinese Hong Kong residents who are able to communicate in Cantonese or Mandarin;
* A current clinical Diagnostic and Statistical Manual of Mental Disorders-fifth edition (DSM-5) diagnosis of insomnia disorder (Primary in nature) according to the Brief Insomnia Questionnaire (BIQ), a validated diagnostic tool. The criteria include having difficulties in falling asleep, difficulties in staying asleep, or early morning awakening with clinically significant consequences for daily life for at least 3 months;
* Insomnia Severity Index total score of at least 10 indicating insomnia at the clinical level;
* Willing to give informed consent and comply with the trial protocol;
* Ambulant and independent in activities of daily living;
* Physically inactive which refers to less than 150 minutes moderate-intensity activity per week or less than 75 minutes vigorous-intensity activity per week, or an equivalent combination of moderate- and vigorous- intensity activity.

Exclusion Criteria:

* Evidence of association of insomnia with medical conditions, other sleep disorders, or side-effects of medications;
* Use of medication or psychotherapeutic components for insomnia or other psychiatric disorders;
* Other possible psychiatric disorders including generalized anxiety disorder (GAD), major depressive disorder (MDD), posttraumatic stress disorder (PTSD), psychosis as screened by structural clinical interview of DSM-IV;
* cognitive impairment preventing informed consent or understanding of instructions (score < 22 in Montreal Cognitive Assessment Hong Kong version);
* Shift work;
* body mass index equal to or over 27.5, the obese criteria for Asians;
* Unsafe conditions or incapable to exercise as recommended by their physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | week 8
  The subjects rate the severity of insomnia, the distress, and the functional impairment associated with insomnia on a 5-point

SECONDARY OUTCOMES:
Sleep diary (7-day) | Baseline, week 4, week 8
  The standardized sleep diary records the daily bedtime and rising time, from which the total time in bed (TIB) can be calculated.
Multidimensional fatigue inventory-20 | Baseline, week 4, week 8
  Multidimensional fatigue inventory-20 is a 20-items self-report instrument designed to measure severity of fatigue.
Hospital Anxiety and Depression Scale | Baseline, week 4, week 8
  The Hospital Anxiety and Depression Scale is a 14-items self-administered questionnaire, which assesses the severity of depressive and anxiety symptoms
Actigraphy (7-day) | Baseline, week 8
  Actigraphy measures wrist movements to assess sleep or waking state, is accomplished through an accelerometer in a wrist worn device
Short Form-6 Dimension | Baseline, week 4, week 8
  The Short Form-6 Dimension is composed of six multi-level dimensions to assess the quality of life which can be used in cost-utility analysis.
Hand grip strength | Baseline, week 8
  Objective hand grip strength
Level of activity | Baseline, week4, week 8
  Self-report level of activity in moderate and vigorous intensity
Weight | Baseline, week 8
  Weight in kilograms; (Weight and Height will be combined to report as BMI in kg/m^2)
Height | Baseline, week 8
  Height in meters; (Weight and Height will be combined to report as BMI in kg/m^2)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, the Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeung WF, Lai AY, Ho FY, Suen LK, Chung KF, Ho JY, Ho LM, Yu BY, Chan LY, Lam TH. Effects of Zero-time Exercise on inactive adults with insomnia disorder: a pilot randomized controlled trial. Sleep Med. 2018 Dec;52:118-127. doi: 10.1016/j.sleep.2018.07.025. Epub 2018 Aug 24. PMID 30312957